CLINICAL TRIAL: NCT01390441
Title: A Two-Part, Phase I Randomized, Double-Blind, Active-Comparator Controlled, Parallel Group Study to Assess the Pharmacokinetics, Safety, and Tolerability of MK-8808 and to Compare the Pharmacokinetics of MK-8808 With EU-approved MabThera® and US-licensed Rituxan® in Patients With Rheumatoid Arthritis (RA)
Brief Title: A Study of the Pharmacokinetics and Safety of MK-8808 (MK-8808-002)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated early by the Sponsor for business reasons.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8808-002
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Results first posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; RA; Rituximab; Rituxan; MabThera; Methotrexate; Rheumatrex; Trexall; MK-8808
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; Methotrexate; Methylprednisolone; Acetaminophen; Loratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part A: MK-8808 500 mg/m^2 / Extension A: MK-8808 1000 mg (Experimental): During the Treatment Period, participants receive one course of MK-8808 (500 mg/m^2) administered intravenously (IV) on Day 1 and Day 15 (with a second optional course of treatment at Weeks 26 and 28). Participants are followed up to Week 52 in the Treatment Period.
  During the Extension Period, participants receive open-label MK-8808 (1000 mg) administered IV at Week 54 and Week 56 (with a second optional course at Weeks 80 and 82). Participants are followed up to Week 106 in the Extension Period.
  Methotrexate 12.5 to 25 mg/week is administered either orally, subcutaneously (SC), or intramuscularly (IM) for the duration of the trial. A 10 mg dose may be administered if a greater dose is not tolerated.
  Interventions: Biological: MK-8808; Drug: Methotrexate; Drug: Methylprednisolone; Drug: Acetaminophen; Drug: Loratadine
- Part A: MabThera® 500 mg/m^2 / Extension A: MK-8808 1000 mg (Active Comparator): During the Treatment Period, participants receive one course of MabThera® (500 mg/m^2) administered IV on Day 1 and Day 15 (with a second optional course of treatment at Weeks 26 and 28). Participants are followed up to Week 52 in the Treatment Period.
  During the Extension Period, participants receive open label MK-8808 (1000 mg) administered IV at Week 54 and Week 56 (with a second optional course at Weeks 80 and 82). Participants are followed up to Week 106 in the Extension Period.
  Methotrexate 12.5 to 25 mg/week is administered either orally, SC, or IM for the duration of the trial. A 10 mg dose may be administered if a greater dose is not tolerated.
  Interventions: Biological: MK-8808; Biological: MabThera® (rituximab); Drug: Methotrexate; Drug: Methylprednisolone; Drug: Acetaminophen; Drug: Loratadine
- Part B: MK-8808 1000 mg / Extension B: MK-8808 1000 mg (Experimental): In the Treatment Period, participants receive one course of MK-8808 (1000 mg) administered IV on Day 1 and Day 15 (with a second optional course of treatment at Weeks 26 and 28). Participants are followed up to Week 52 in the Treatment Period.
  In the Extension Period, participants receive open label MK-8808 (1000 mg) adminstered IV at Week 54 and Week 56 (with a second optional course at Weeks 80 and 82). Participants are followed up to Week 106 in the Extension Period.
  Methotrexate 12.5 to 25 mg/week is administered either orally, SC, or IM for the duration of the trial. A 10 mg dose may be administered if a greater dose is not tolerated.
  Interventions: Biological: MK-8808; Drug: Methotrexate; Drug: Methylprednisolone; Drug: Acetaminophen; Drug: Loratadine
- Part B: MabThera® 1000 mg / Extension B: MK-8808 1000 mg (Active Comparator): In the Treatment Period, participants receive one course of MabThera® (1000 mg) administered IV on Day 1 and Day 15 (with a second optional course of treatment at Weeks 26 and 28). Participants are followed up to Week 52 in the Treatment Period.
  In the Extension Period, participants receive open label MK-8808 (1000 mg) administered IV at Week 54 and Week 56 (with a second optional course at Weeks 80 and 82). Participants are followed up to Week 106 in the Extension Period.
  Methotrexate 12.5 to 25 mg/week is administered either orally, SC, or IM for the duration of the trial. A 10 mg dose may be administered if a greater dose is not tolerated.
  Interventions: Biological: MK-8808; Biological: MabThera® (rituximab); Drug: Methotrexate; Drug: Methylprednisolone; Drug: Acetaminophen; Drug: Loratadine
- Part B: Rituxan® 1000 mg / Extension B: MK-8808 1000 mg (Experimental): In the Treatment Period, participants receive one course of Rituxan® (1000 mg) administered IV on Day 1 and Day 15 (with a second optional course of treatment at Weeks 26 and 28). Participants are followed up to Week 52 in the Treatment Period.
  In the Extension Period, participants receive open label MK-8808 (1000 mg) administered IV at Week 54 and Week 56 (with a second optional course at Weeks 80 and 82). Participants are followed up to Week 106 in the Extension Period.
  Methotrexate 12.5 to 25 mg/week is administered either orally, SC, or IM for the duration of the trial. A 10 mg dose may be administered if a greater dose is not tolerated.
  Interventions: Biological: MK-8808; Drug: Methotrexate; Biological: Rituxan® (rituximab); Drug: Methylprednisolone; Drug: Acetaminophen; Drug: Loratadine

INTERVENTIONS:
Biological: MK-8808 — MK-8808 500 mg/m^2 administered by IV on Day 1 and Day 15 or MK-8808 1000 mg administered by IV at Week 54 and Week 56
Biological: MabThera® (rituximab) — MabThera® 500 mg/m^2 or 1000 mg administered by IV on Day 1 and Day 15
  Other Names: Rituxan®; Rituximab
  Arms: Part A: MabThera® 500 mg/m^2 / Extension A: MK-8808 1000 mg; Part B: MabThera® 1000 mg / Extension B: MK-8808 1000 mg
Drug: Methotrexate — Methotrexate 10-25 mg administered orally, SC, or IM as a weekly stable dose
  Other Names: Trexall®; Rheumatrex®
Biological: Rituxan® (rituximab) — Rituxan® 1000 mg administered by IV on Day 1 and Day 15
  Other Names: Rituximab
  Arms: Part B: Rituxan® 1000 mg / Extension B: MK-8808 1000 mg
Drug: Methylprednisolone — Methylprednisolone 100 mg administered IV before initiation of each infusion as pre-medication to reduce the incidence and severity of infusion reactions
Drug: Acetaminophen — Acetaminophen 1000 to 1350 mg administered orally before initiation of each infusion as pre-medication to reduce the incidence and severity of infusion reactions
  Other Names: Paracetamol
Drug: Loratadine — Loratidine 10 mg administered orally before initiation of each infusion as pre-medication to reduce the incidence and severity of infusion reactions
  Other Names: Claritin®

SUMMARY:
This is a study of the overall safety, tolerability, and pharmacokinetics (PK) of MK-8808 versus rituximab (MabThera® and Rituxan®) in participants with moderate to severe RA with an inadequate response or intolerance to methotrexate.

DETAILED DESCRIPTION:
In Part A of the base study, participants are randomized to either MK-8808 or MabThera®. In Part B of the base study, participants are randomized to either MK-8808, MabThera®, or Rituxan®. Participants enrolled in Part A are not eligible to participate in Part B. In both Parts A and B, participants will receive one or two courses of therapy, with each course including two infusions of the study drugs.

The extension portion of the study (Part C) will sequentially follow the base study beginning at Week 52 and continue for an additional 54 weeks. All participants who meet eligibility criteria and continue into the study extension will be treated with open-label MK-8808. Participants randomized to MK-8808 in the base study will remain on the same therapy. Participants randomized to rituximab (MabThera® or Rituxan®) in the base study will be switched to MK-8808 for the extension study.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of reproductive potential must demonstrate a serum β-human chorionic gonadotropin (hCG) level consistent with the nongravid state at the pre-study (screening) visit, and a negative urine pregnancy test within 24 hours prior to all doses and agree to use (and/or have their partner use) two acceptable methods of birth control beginning at least 2 weeks prior to administration of the first dose of study drug, throughout the study (including washout intervals between treatment periods/panels) and until at least 12 months after administration of the last dose of study drug in the last treatment period
* The participant has a Body Mass Index (BMI) ≤35 kg/m^2 at the prestudy (screening) visit
* For Part A Only: The participant has a body surface are (BSA) ≤2.0 m^2 at the prestudy (screening) visit.
* Has satisfied at least 4 of 7 American Rheumatology Association (ARA) 1987 revised criteria for the diagnosis of RA
* Is American College of Rheumatology (ACR) Functional Class I, II, or III
* Had a diagnosis of RA made at least 6 months prior to the prestudy (screening) visit, was ≥ 16 years of age when diagnosed, and has active disease
* Is on a stable oral, IM, or SC dose of methotrexate and is continuing to take methotrexate
* Has an inadequate response or intolerance to at least one disease-modifying antirheumatic drug (DMARD)
* For Part A: Participant is either naïve to biological therapy for RA or has had an inadequate response to previous or current treatment with an anti-tumor necrosis factor (TNF) treatment (patient could have failed up to three anti-TNF agents treatments) or participant has had intolerance up to three anti-TNF treatments.
* For Part B: Participant has had an inadequate response to previous or current treatment with an anti-TNF treatment (patient could have failed up to three anti-TNF agents treatments) or participant has had intolerance up to three anti-TNF treatments
* Participant has no clinically significant abnormality on electrocardiogram performed at the prestudy (screening) visit and/or prior to administration of the initial dose of study drug
* For Part B Only: Participant is positive for rheumatoid factor (RF) or, if negative for RF, is positive for anti-CCP at screening visit
* For Part C Only: Participant must have completed the first 52 weeks of treatment in the base study
* For Part C Only: Participant achieved a minimum 20% response from baseline on the American College of Rheumatology (ACR) Responder Index (ACR20) at Visit 19 (last visit for the base study)

Exclusion Criteria:

* Mentally or legally incapacitated, has significant emotional problems at the time of the prestudy (screening) visit or during the conduct of the study or has a history of a clinically significant psychiatric disorder over the last 5 years
* Creatinine clearance of ≤ 80 mL/min
* History of stroke, chronic seizures or major neurological disorder
* History of neoplastic disease, except treated basal cell carcinoma or carcinoma in situ of the cervix or other malignancies which have been successfully treated ≥ 5 years
* History of leukemia, lymphoma, malignant melanoma, or myeloproliferative disease regardless of the time since treatment
* History of coronary artery disease, congestive heart failure (New York Heart Association Class I-IV), or a history of clinically significant arrhythmia (including any history of atrial fibrillation, atrial flutter, or any sustained ventricular arrhythmia)
* Hypersensitivity or allergy to rituximab or any of the excipients of MK-8808 or rituximab (MabThera® or Rituxan® )
* History of a rheumatic autoimmune disease other than RA (e.g. systemic lupus erythematosus (SLE), polymyositis, etc.)
* Severe active infection of any type or history of a medically serious infection as defined by a history of treatment requiring hospitalization, long term IV outpatient treatment for systemic bacterial, viral or fungal infection, use of IV antibiotics within 30-days of screening, or use of antibiotic therapy three or more times in the last six months prior to screening
* History of opportunistic infection
* Active-virus vaccination within 4 weeks
* Active tuberculosis with or without adequate treatment, history of latent tuberculosis without written confirmation from health care provider of adequate prophylaxis or any evidence of tuberculosis on a chest X-ray performed within 3 months of dosing
* Chronic hepatitis B or hepatitis C infection or has human immunodeficiency virus (HIV) infection
* Previously treated with rituximab (MabThera® or Rituxan®) or any investigational anti-CD20 antibody
* Active use or planned use of a prohibited DMARD during the course of study participation, and/or insufficient washout from a prohibited DMARD at the time of the planned first dose of MK-8808/rituximab (MabThera® or Rituxan®)
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks
* Participated in another investigational study with length of time within at least 5 half-lives of the previous investigational study drug
* Pregnant or breastfeeding or expecting to conceive
* Allergy to murine proteins
* Allergy or sensitivity to components of the drug vial or any of the materials used for infusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled participants 18 to 65 years of age with a diagnosis of moderate/severe rheumatoid arthritis (RA), naive to treatment or having failed >=1 anti-TNF agent, and on a stable dose of methotrexate. Not all participants completing the Treatment Period entered the Extension Period due to study early termination.
Pre-assignment Details: For Part B only, positive for rheumatoid factor (RF) or, if negative for RF, positive for anti-cyclic citrullinated protein antibodies at the screening visit.
Groups:
- Part A: MK-8808 500 mg/m^2 / Extension A: MK-8808 1000 mg: Participants receive one course of MK-8808 (500 mg/m^2) administered intravenously (IV) on Day 1 and Day 15 (2nd optional course of treatment at Weeks 26 and 28) in the Treatment Period (up to Week 52) followed by open-label MK-8808 (1000 mg) IV at Week 54 and Week 56 (2nd optional course at Weeks 80 and 82) in the Extension Period (up to Week 106) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, subcutaneously (SC), or intramuscularly (IM) for the duration of the trial.
- Part A: MabThera® 500 mg/m^2 / Extension A: MK-8808 1000 mg: Participants receive one course of MabThera® (500 mg/m^2) administered IV on Day 1 and Day 15 (2nd optional course of treatment at Weeks 26 and 28) in the Treatment Period (up to Week 52) followed by open label MK-8808 1000 mg IV at Week 54 and Week 56 (2nd optional course at Weeks 80 and 82) in the Extension Period (up to Week 106) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
- Part B: MK-8808 1000 mg / Extension B: MK-8808 1000 mg: Participants receive one course of MK-8808 (1000 mg) IV on Day 1 and Day 15 (2nd optional course of treatment at Weeks 26 and 28) in the Treatment Period (up to Week 52) followed by open label MK-8808 1000 mg IV at Week 54 and Week 56 (2nd optional course at Weeks 80 and 82) in the Extension Period (up to Week 106) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
- Part B: MabThera® 1000 mg / Extension B: MK-8808 1000 mg: Participants receive one course of MabThera® (1000 mg) IV on Day 1 and Day 15 (2nd optional course of treatment at Weeks 26 and 28) in the Treatment Period (up to Week 52) followed by open label MK-8808 1000 mg IV at Week 54 and Week 56 (2nd optional course at Weeks 80 and 82) in the Extension Period (up to Week 106) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
- Part B: Rituxan® 1000 mg / Extension B: MK-8808 1000 mg: Participants receive one course of Rituxan® (1000 mg) administered IV on Day 1 and Day 15 (2nd optional course of treatment at Weeks 26 and 28) in the Treatment Period (up to Week 52) followed by open label MK-8808 1000 mg IV at Week 54 and Week 56 (2nd optional course at Weeks 80 and 82) in the Extension Period (up to Week 106) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
Period: Treatment Period
Arm/Group | Part A: MK-8808 500 mg/m^2 / Extension A: MK-8808 1000 mg | Part A: MabThera® 500 mg/m^2 / Extension A: MK-8808 1000 mg | Part B: MK-8808 1000 mg / Extension B: MK-8808 1000 mg | Part B: MabThera® 1000 mg / Extension B: MK-8808 1000 mg | Part B: Rituxan® 1000 mg / Extension B: MK-8808 1000 mg
Started | 23 | 22 | 18 | 19 | 18
Completed | 22 | 21 | 8 | 6 | 7
Not Completed | 1 | 1 | 10 | 13 | 11
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1
Not completed — Unknown due to early stopping of study | 0 | 0 | 8 | 11 | 7
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Period: Extension Period
Arm/Group | Part A: MK-8808 500 mg/m^2 / Extension A: MK-8808 1000 mg | Part A: MabThera® 500 mg/m^2 / Extension A: MK-8808 1000 mg | Part B: MK-8808 1000 mg / Extension B: MK-8808 1000 mg | Part B: MabThera® 1000 mg / Extension B: MK-8808 1000 mg | Part B: Rituxan® 1000 mg / Extension B: MK-8808 1000 mg
Started | 15 (Not all participants entered the Extension Period due to early termination of the study.) | 13 (Not all participants entered the Extension Period due to early termination of the study.) | 1 (Not all participants entered the Extension Period due to early termination of the study.) | 1 (Not all participants entered the Extension Period due to early termination of the study.) | 3 (Not all participants entered the Extension Period due to early termination of the study.)
Completed | 12 | 12 | 1 | 0 | 3
Not Completed | 3 | 1 | 0 | 1 | 0
Not completed — Protocol Violation | 3 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A: MK-8808 500 mg/m^2: Participants receive one course of MK-8808 (500 mg/m^2) administered intravenously (IV) on Day 1 and Day 15; (2nd optional course of treatment at Weeks 26 and 28) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
- Part A: MabThera® 500 mg/m^2: Participants receive one course of MabThera® (500 mg/m^2) administered IV on Day 1 and Day 15 (2nd optional course of treatment at Weeks 26 and 28) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
- Part B: MK-8808 1000 mg: Participants receive one course of MK-8808 (1000 mg) IV on Day 1 and Day 15 (2nd optional course of treatment at Weeks 26 and 28) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
- Part B: MabThera® 1000 mg: Participants receive one course of MabThera® (1000 mg) IV on Day 1 and Day 15 (2nd optional course of treatment at Weeks 26 and 28) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
- Part B: Rituxan® 1000 mg: Participants receive one course of Rituxan® (1000 mg) administered IV on Day 1 and Day 15 (2nd optional course of treatment at Weeks 26 and 28) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
- Total: Total of all reporting groups
Arm/Group | Part A: MK-8808 500 mg/m^2 | Part A: MabThera® 500 mg/m^2 | Part B: MK-8808 1000 mg | Part B: MabThera® 1000 mg | Part B: Rituxan® 1000 mg | Total
Number analyzed (Participants) | 23 | 22 | 18 | 19 | 18 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (6.7) | 51.5 (8.4) | 46.4 (10.9) | 48.7 (12.4) | 46.2 (10.5) | 49.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 14 | 16 | 15 | 84
  Male | 3 | 3 | 4 | 3 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Part A: Area Under the Concentration-time Curve From Day 0 to Day 84 (AUC0-84day) After a Single Course of Treatment
Description: AUC is a measure of the amount of drug in the plasma over time; samples are collected at intervals from pre-dose up to 84 days after the dose. Descriptive data values and associated dispersion measures (confidence intervals) are expressed in terms of the factor 10E6.
Time Frame: Day 1 (pre- and post-dose), Day 3, Day 5, Day 8, Day 15, Day 17, Day 19, Day 22, Day 29, Day 43, Day 57, Day 85
Population: Participants who completed a full course of MK-8808 or MabThera® (two full doses of 500 mg/m^2 on Days 1 and 15), had no major protocol violations, had a complete pharmacokinetic (PK) profile, had serum MK-8808 or MabThera® concentrations prior to the first dose of the first course not exceeding 5% of Cmax after the first dose of the first course
Measure: Geometric Mean (95% Confidence Interval); unit: hr*mg/mL
Groups:
- Part A: MK-8808 500 mg/m^2: Participants receive one course of MK-8808 (500 mg/m^2) administered IV on Day 1 and Day 15 (2nd optional course of treatment at Weeks 26 and 28) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
Arm/Group | Part A: MK-8808 500 mg/m^2 | Part A: MabThera® 500 mg/m^2
Number analyzed (Participants) | 22 | 19
hr*mg/mL | 110.56 [94.51 to 129.32] | 110.12 [91.97 to 131.84]
Statistical Analysis 1: Comparison: Part A: MK-8808 500 mg/m^2 vs Part A: MabThera® 500 mg/m^2; Back-transformed least squares mean and confidence interval from fixed effects model performed on natural log-transformed values containing treatment as a fixed effect and gender as a covariate; Test type: Non-Inferiority or Equivalence — PK bioequivalence was assumed if the 90% confidence interval of the geometric mean ratio for the comparison fell within the range 0.80-1.25; ANOVA; Geometric mean ratio = 1.00, 90% CI 2-sided [0.87 to 1.16]

2. Primary Outcome: Part B: Area Under the Concentration-time Curve From Day 0 to Day 84 (AUC0-84day) After a Single Course of Treatment
Description: AUC is a measure of the amount of drug in the plasma over time; samples are collected at intervals from pre-dose up to 84 days after the dose.
Time Frame: Day 1 (pre- and post-dose), Day 3, Day 5, Day 8, Day 15, Day 17, Day 19, Day 22, Day 29, Day 43, Day 57, Day 85
Population: PK analysis for Part B was not performed due to early termination of the study after Part A. Blood sampling in Part B was performed without further laboratory quantification for this outcome measure.
Arm/Group | Part B: MK-8808 1000 mg | Part B: MabThera® 1000 mg | Part B: Rituxan® 1000 mg
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event
Description: An adverse event is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure.
Time Frame: Parts A and B: Up to 52 weeks; Extension A and B: Up to 106 weeks
Population: All Participants as Treated (APaT) population defined as all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Groups:
- Part A: MabThera 500 mg/m^2: Participants receive one course of MabThera® (500 mg/m^2) administered IV on Day 1 and Day 15 (2nd optional course of treatment at Weeks 26 and 28) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
- Part B: MabThera 1000 mg: Participants receive one course of MabThera (1000 mg) IV on Day 1 and Day 15 (2nd optional course of treatment at Weeks 26 and 28) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
- Part B: Rituxan 1000 mg: Participants receive one course of Rituxan (1000 mg) administered IV on Day 1 and Day 15 (2nd optional course of treatment at Weeks 26 and 28) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
- Extension A: MK-8808 500 mg/m^2 /MK-8808 1000 mg: Participants who completed Part A MK-8808 500 mg/m^2 therapy will receive open-label MK-8808 (1000 mg) IV at Week 54 and Week 56 (2nd optional course at Weeks 80 and 82) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
- Extension A: MabThera 500 mg/m^2 /MK-8808 1000 mg: Participants who completed Part A MabThera therapy will receive open label MK-8808 1000 mg IV at Week 54 and Week 56 (2nd optional course at Weeks 80 and 82) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
- Extension B: MK-8808 1000 mg /MK-8808 1000 mg: Participants who completed Part B MK-8808 will receive open label MK-8808 1000 mg IV at Week 54 and Week 56 (2nd optional course at Weeks 80 and 82) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
- Extension B: MabThera 1000 mg /MK-8808 1000 mg: Participants who completed Part B MabThera will receive open label MK-8808 1000 mg IV at Week 54 and Week 56 (2nd optional course at Weeks 80 and 82) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
- Extension B: Rituxan1000 mg/MK-8808 1000 mg: Participants who completed Part B Rituxan will receive open label MK-8808 1000 mg IV at Week 54 and Week 56 (2nd optional course at Weeks 80 and 82) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
Arm/Group | Part A: MK-8808 500 mg/m^2 | Part A: MabThera 500 mg/m^2 | Part B: MK-8808 1000 mg | Part B: MabThera 1000 mg | Part B: Rituxan 1000 mg | Extension A: MK-8808 500 mg/m^2 /MK-8808 1000 mg | Extension A: MabThera 500 mg/m^2 /MK-8808 1000 mg | Extension B: MK-8808 1000 mg /MK-8808 1000 mg | Extension B: MabThera 1000 mg /MK-8808 1000 mg | Extension B: Rituxan1000 mg/MK-8808 1000 mg
Number analyzed (Participants) | 23 | 22 | 18 | 19 | 18 | 15 | 13 | 1 | 1 | 3
Participants | 18 | 21 | 12 | 16 | 13 | 2 | 2 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Part A: MK-8808 500 mg/m^2 vs Part A: MabThera 500 mg/m^2; The difference in percent AE incidence was determined for the treatment comparison (Part A: MK-8808 500 mg/m^2 - Part A: MabThera 500 mg/m^2) when >=4 participants in an arm experienced an event; Test type: Superiority or Other; Miettinen-Nurminen; Percent difference = -17.2, 95% CI 2-sided [-38.6 to 3.6]
Statistical Analysis 2: Comparison: Part B: MK-8808 1000 mg vs Part B: MabThera 1000 mg; The difference in percent AE incidence was determined for the treatment comparison (Part B: MK-8808 1000 mg - Part B: MabThera 1000 mg) when >=4 participants in an arm experienced an event; Test type: Superiority or Other; Miettinen-Nurminen; Percent difference = -17.5, 95% CI 2-sided [-44.4 to 10.9]
Statistical Analysis 3: Comparison: Part B: MK-8808 1000 mg vs Part B: Rituxan 1000 mg; The difference in percent AE incidence was determined for the treatment comparison (Part B: MK-8808 1000 mg - Part B: Rituxan® 1000 mg) when >=4 participants in an arm experienced an event; Test type: Superiority or Other; Miettinen-Nurminen; Percent difference = -5.6, 95% CI 2-sided [-34.9 to 24.6]
Statistical Analysis 4: Comparison: Part B: MabThera 1000 mg vs Part B: Rituxan 1000 mg; The difference in percent AE incidence was determined for the treatment comparison (Part B: MabThera® 1000 mg - Part B: Rituxan® 1000 mg) when >=4 participants in an arm experienced an event; Test type: Superiority or Other; Miettinen-Nurminen; Percent differnce = 12.0, 95% CI 2-sided [-15.6 to 38.9]

4. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to Adverse Events
Description: Discontinuation/withdrawal of study treatment due to an adverse event was performed at the discretion of the investigator or the Sponsor for safety concerns. An adverse event is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure.
Time Frame: Parts A and B: Up to Week 28; Extension A and B: Up to 82 weeks
Population: APaT population defined as all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Groups:
- Extension A: MabThera® 500 mg/m^2 /MK-8808 1000 mg: Participants who completed Part A MabThera® therapy will receive open label MK-8808 1000 mg IV at Week 54 and Week 56 (2nd optional course at Weeks 80 and 82) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
- Extension B: MabThera® 1000 mg /MK-8808 1000 mg: Participants who completed Part B MabThera® will receive open label MK-8808 1000 mg IV at Week 54 and Week 56 (2nd optional course at Weeks 80 and 82) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
- Extension B: Rituxan® 1000 mg/MK-8808 1000 mg: Participants who completed Part B Rituxan® will receive open label MK-8808 1000 mg IV at Week 54 and Week 56 (2nd optional course at Weeks 80 and 82) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
Arm/Group | Part A: MK-8808 500 mg/m^2 | Part A: MabThera® 500 mg/m^2 | Part B: MK-8808 1000 mg | Part B: MabThera® 1000 mg | Part B: Rituxan® 1000 mg | Extension A: MK-8808 500 mg/m^2 /MK-8808 1000 mg | Extension A: MabThera® 500 mg/m^2 /MK-8808 1000 mg | Extension B: MK-8808 1000 mg /MK-8808 1000 mg | Extension B: MabThera® 1000 mg /MK-8808 1000 mg | Extension B: Rituxan® 1000 mg/MK-8808 1000 mg
Number analyzed (Participants) | 23 | 22 | 18 | 19 | 18 | 15 | 13 | 1 | 1 | 3
Participants | 2 | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Part A: Maximum Concentration (Cmax) After the Second Infusion of a Single Course of Treatment
Description: Cmax is a measure of the maximum plasma concentration of drug; samples are collected on Day 15 after the second infusion of the first course of treatment. Descriptive data values and associated dispersion measures (confidence intervals) are expressed in terms of the factor 10E3.
Time Frame: Day 15
Population: Participants who completed a full course of MK-8808 or MabThera® (two full doses of 500 mg/m^2 on Days 1 and 15); had no major protocol violations; had a complete PK profile; had serum MK-8808 or MabThera® concentrations prior to the first dose of the first course not exceeding 5% of Cmax after the first dose of the first course.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Part A: MK-8808 500 mg/m^2 | Part A: MabThera® 500 mg/m^2
Number analyzed (Participants) | 22 | 19
ng/mL | 326.49 [287.72 to 370.49] | 332.39 [287.48 to 384.31]
Statistical Analysis 1: Comparison: Part A: MK-8808 500 mg/m^2 vs Part A: MabThera® 500 mg/m^2; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Geometric mean ratio = 0.98, 90% CI 2-sided [0.87 to 1.1]

6. Secondary Outcome: Part B: Cmax After the Second Infusion of a Single Course of Treatment
Description: Cmax is a measure of the maximum plasma concentration of drug; samples are collected on Day 15 after the second infusion of the first course of treatment.
Time Frame: Day 15
Population: as for outcome 2
Arm/Group | Part B: MK-8808 1000 mg | Part B: MabThera® 1000 mg | Part B: Rituxan® 1000 mg
Number analyzed (Participants) | 0 | 0 | 0

7. Other Pre Specified Outcome: Part A: Number of ACR20, ACR50, and ACR70 Responders at Week 24
Description: American College of Rheumatology (ACR) Responder Index is based on a set of evaluations: the Investigator Tender Joint Count/Number of Tender Joints (out of 68 Joints); Investigator Swollen Joint Count/Number of Swollen Joints (out of 66 Joints); Patient Global Assessment of Disease Activity (PGAD); Investigator Global Assessment of Disease Activity (IGAD); Patient Global Assessment of Pain (PGAP); Health Assessment Questionnaire Disability Index (HAQ-DI); and ESR. ACR response indicates percent change (ie, improvement) from baseline (20%, 50%, 70%) PGAD & IGAD: assessment of function on a 4-point Likert scale: 0=very well to 3=unable to do PGAP: pain due to arthritis measured on a 0-100 mm visual analog scale: Left hand marker-"no pain"; right hand marker-"extreme pain" HAQ-DI: assessment of 8 daily living activities (dress/groom; arise; eat; walk; reach; grip; hygiene; common daily activities) on 4-point Likert scale: 0=no difficulty to 3=unable to do
Time Frame: Week 24
Population: Full Analysis Set defined as all randomized participants who received at least one complete treatment course (2 doses) and had at least one post-treatment measurement. Patients were included in the treatment group to which they were randomized. A patient might have been be excluded from the FAS population for a given endpoint for multiple reasons.
Measure: Number; unit: Participants
Groups:
- Part A: MK-8808 500 mg/m^2: Participants receive one course of MK-8808 (500 mg/m^2) administered IV on Day 1 and Day 15 (2nd optional course of treatment at Weeks 26 and 28) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, subcutaneously SC, or IM for the duration of the trial.
Arm/Group | Part A: MK-8808 500 mg/m^2 | Part A: MabThera® 500 mg/m^2
Number analyzed (Participants) | 23 | 21
Participants
  ACR20 | 23 | 20
  ACR50 | 16 | 15
  ACR70 | 4 | 4

8. Other Pre Specified Outcome: Part B: Number of ACR20, ACR50, and ACR70 Responders at Week 24
Description: as for outcome 7
Time Frame: Week 24
Population: FAS defined as all randomized participants who received at least one complete treatment course (2 doses) and had at least one post-treatment measurement. Patients were included in the treatment group to which they were randomized. A patient might have been be excluded from the FAS population for a given endpoint for multiple reasons.
Measure: Number; unit: Participants
Arm/Group | Part B: MK-8808 1000 mg | Part B: MabThera® 1000 mg | Part B: Rituxan® 1000 mg
Number analyzed (Participants) | 17 | 18 | 17
Participants
  ACR20 | 16 | 17 | 15
  ACR50 | 12 | 12 | 13
  ACR70 | 2 | 1 | 1

9. Other Pre Specified Outcome: Change From Baseline in Disease Activity in 28 Joints C-Reactive Protein Score (DAS28-CRP) by Time-point
Description: The DAS28-CRP is a combination scoring method for function using the European League against Rheumatism (EULAR) 28 joint count and the CRP value. The DAS28-CRP scores range from 2.0 to 10.0 with higher values indicating a higher disease activity. A DAS28-CRP below the score of 2.6 is interpreted as Remission. CRP values below lower limit of quantification (LLQ) (<0.4 mg/dL) were set to 0.2 mg/dL in the calculation of DAS28-CRP.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score
Groups:
- Part A: MK-8808 500 mg/m^2: Participants receive one course of MK-8808 (500 mg/m^2) administered IV on Day 1 and Day 15 (2nd optional course of treatment at Weeks 26 and 28) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, subcutaneously (SC), or IM for the duration of the trial.
Arm/Group | Part A: MK-8808 500 mg/m^2 | Part A: MabThera® 500 mg/m^2
Number analyzed (Participants) | 23 | 21
Score
  Week 6 (n=22, n=20) | -1.39 (1.02) | -1.16 (1.26)
  Week 12 (n=21, n=21) | -1.68 (1.12) | -2.04 (1.39)
Statistical Analysis 1: Comparison: Part A: MK-8808 500 mg/m^2 vs Part A: MabThera® 500 mg/m^2; Estimated difference vs MabThera® at 6 weeks; Test type: Non-Inferiority or Equivalence; ANCOVA; The model included a term for treatment; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.9 to 0.5]
Statistical Analysis 2: Comparison: Part A: MK-8808 500 mg/m^2 vs Part A: MabThera® 500 mg/m^2; Estimated difference vs MabThera® at 12 weeks; Test type: Non-Inferiority or Equivalence; ANCOVA; The model included a term for treatment; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.4 to 1.2]

10. Primary Outcome: Number of Participants With Immunoglobulin G (IgG) Response in the Extension Study
Description: Serum IgG levels are determined over course of therapy with MK-8808 in the Extension Study.
Time Frame: Week 54, Week 68, Week 80, Week 94, Week 106
Population: The analysis was not performed due to early termination of the study after Part A. Blood sampling in the Extension Study was performed without further laboratory quantification for this outcome measure.
Arm/Group | Extension A: MK-8808 500 mg/m^2 /MK-8808 1000 mg | Extension A: MabThera® 500 mg/m^2 /MK-8808 1000 mg | Extension B: MK-8808 1000 mg /MK-8808 1000 mg | Extension B: MabThera® 1000 mg /MK-8808 1000 mg | Extension B: Rituxan® 1000 mg/MK-8808 1000 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Participants Positive for Anti-Drug Antibody (ADA) Formation in the Extension Study
Description: Serum ADA positivity is determined over course of therapy with MK-8808 in the Extension Study.
Time Frame: Week 54, Week 56, Week 68, Week 80, Week 82, Week 94, Week 106
Population: as for outcome 10
Arm/Group | Extension A: MK-8808 500 mg/m^2 /MK-8808 1000 mg | Extension A: MabThera® 500 mg/m^2 /MK-8808 1000 mg | Extension B: MK-8808 1000 mg /MK-8808 1000 mg | Extension B: MabThera® 1000 mg /MK-8808 1000 mg | Extension B: Rituxan® 1000 mg/MK-8808 1000 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Parts A and B: Up to 52 weeks; Extension A and B: Up to 106 weeks
Description: An adverse event is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure. The APaT population was used for safety analysis.
Groups:
- Part A: MK-8808 500 mg/m^2: Participants receive one course of MK-8808 (500 mg/m^2) administered IV on Day 1 and Day 15; (2nd optional course of treatment at Weeks 26 and 28) + methotrexate 12.5 to 25 mg/week (or 10 mg if greater dose not tolerated) either orally, SC, or IM for the duration of the trial.
Arm/Group | Part A: MK-8808 500 mg/m^2 | Part A: MabThera 500 mg/m^2 | Part B: MK-8808 1000 mg | Part B: MabThera 1000 mg | Part B: Rituxan 1000 mg | Extension A: MK-8808 500 mg/m^2 /MK-8808 1000 mg | Extension A: MabThera® 500 mg/m^2 /MK-8808 1000 mg | Extension B: MK-8808 1000 mg /MK-8808 1000 mg | Extension B: MabThera® 1000 mg /MK-8808 1000 mg | Extension B: Rituxan® 1000 mg/MK-8808 1000 mg
Serious Adverse Events (participants affected / at risk) | 1/23 | 1/22 | 2/18 | 0/19 | 0/18 | 0/15 | 0/13 | 0/1 | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 15/23 | 17/22 | 11/18 | 16/19 | 13/18 | 2/15 | 2/13 | 0/1 | 0/1 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: MK-8808 500 mg/m^2 (N=23) | Part A: MabThera 500 mg/m^2 (N=22) | Part B: MK-8808 1000 mg (N=18) | Part B: MabThera 1000 mg (N=19) | Part B: Rituxan 1000 mg (N=18) | Extension A: MK-8808 500 mg/m^2 /MK-8808 1000 mg (N=15) | Extension A: MabThera® 500 mg/m^2 /MK-8808 1000 mg (N=13) | Extension B: MK-8808 1000 mg /MK-8808 1000 mg (N=1) | Extension B: MabThera® 1000 mg /MK-8808 1000 mg (N=1) | Extension B: Rituxan® 1000 mg/MK-8808 1000 mg (N=3)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: MK-8808 500 mg/m^2 (N=23) | Part A: MabThera 500 mg/m^2 (N=22) | Part B: MK-8808 1000 mg (N=18) | Part B: MabThera 1000 mg (N=19) | Part B: Rituxan 1000 mg (N=18) | Extension A: MK-8808 500 mg/m^2 /MK-8808 1000 mg (N=15) | Extension A: MabThera® 500 mg/m^2 /MK-8808 1000 mg (N=13) | Extension B: MK-8808 1000 mg /MK-8808 1000 mg (N=1) | Extension B: MabThera® 1000 mg /MK-8808 1000 mg (N=1) | Extension B: Rituxan® 1000 mg/MK-8808 1000 mg (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anisocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercoagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Microcytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polychromasia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis C (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis B surface antigen positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
QRS axis abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cell elliptocytes present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cells urine positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal amyloidosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/ presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.